CLINICAL TRIAL: NCT04759976
Title: Optimize Motor Learning to Improve Neurorehabilitation
Acronym: OnLINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-01179
Record Dates: First submitted 2021-02-01; First posted 2021-02-18 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Neurologic Disorder
Keywords: Neurorehabilitation; Robotic Rehabilitation; Motor Learning
MeSH Terms: conditions — Stroke; Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotic motor training (Experimental): Participants will perform motor tasks (i.e. movements) with upper limb robotic devices applying different strategies (e.g. supporting or challenging the subject, or being fully compliant).
  Interventions: Behavioral: Robotic motor training

INTERVENTIONS:
Behavioral: Robotic motor training — The experiments consist in performing motor tasks with upper-limb robotic devices.

SUMMARY:
The objective of this study is to develop and evaluate novel robotic training strategies that modulate errors based on the subjects' individual motor and cognitive needs. For this purpose, healthy adults and neurologic patients will participate in robotic motor learning experiments. Patients have a diagnosis of a neurological disease (i.e., stroke, spinal cord injury, multiple sclerosis, Guillain-Barré syndrome) limiting arm motor function.

DETAILED DESCRIPTION:
Neurological patients (e.g., after stroke) engage in intensive and expensive neurorehabilitation therapy to regain part of their former motor functional ability to perform everyday activities with often limited and unsatisfactory outcome. Robots became a promising supplement or even alternative for neurorehabilitation therapy, providing cost-effective, high repetition and task-oriented training. However, results of an initial body of work comparing the effectiveness of robotic training strategies are highly inconclusive. A possible explanation is that most current robotic systems cover only one neurorehabilitation strategy (e.g. reducing or augmenting movement errors) and may thus insufficiently address the subjects' individual needs and the characteristics of the task to be learned. In this study, Investigators will perform several motor learning experiments with healthy adult and neurological patients in order to evaluate the relative motor and cognitive benefits of newly developed robotic training strategies that modulate errors based on the subject's age, skill level and tasks characteristics. The effects of the new strategies will be compared to classical robotic assistance, and to non-robotic feedback approaches, such as visual feedback. The culmination of this work may help to optimize training benefits of already existing rehabilitation robots.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Informed Consent as documented by signature ("Informed Consent" form)
* Bodyweight <120 kg
* Ability to communicate effectively with the examiner so that the validity of the patient's data could not be compromised

Exclusion Criteria:

* Excessive spasticity of the affected arm (Ashworth Scale ≥3)
* Serious medical or psychiatric disorder
* Orthopaedic, rheumatological, or other disease restricting movements of the paretic arm
* Shoulder subluxation
* Skin ulcerations at the paretic arm
* Cyber-sickness (i.e., nausea when looking at a screen or playing computer games)
* Serious cognitive defects or aphasia preventing effective use of the robotic devices
* Severe visual and auditory impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Change in kinematic performance assessed by the robot | Baseline, training (immediately after baseline), retention (1-2 days after the training)
  Motion changes from baseline in the kinematic variables assessed by the robot and motion trackers during the motor learning task. The kinematic performance analysis consists of end-effector position in the x, y, and z-axis, in meters, and joint angles in degrees.
Change in kinetic performance assessed by the robot | Baseline, training (immediately after baseline), retention (1-2 days after the training)
  Force changes from baseline in the kinetic variables assessed by the robot using force sensors during the motor learning task. Kinetic performance analysis consists of interaction forces in x, y, and z-axis, in N and applied robot joint torques by the motors, in Nm.
Spatial analysis of changes in evoked potentials as assessed by Electroencephalography (EEG) measurement | Baseline, training (immediately after baseline), retention (1-2 days after the training)
  Electroencephalographical assessment of changes in evoked potentials i.e. the electrical activity of the brain in response to stimulation of specific sensory nerve pathways.

SECONDARY OUTCOMES:
Change in embodiment | Before Intervention, Immediately after the end of intervention
  Virtual Reality (VR) Embodiment Scale, Self administered Likert scale of 1-7 (Strongly Disagree to Strongly Agree)
Spatial analysis of changes in Task-Based Brain Connectivity as assessed by Electroencephalography (EEG) measurement | Baseline, training (immediately after baseline or 1-2 days after baseline), retention (1-2 days after the training)
  Changes in Task-Based Brain Connectivity from baseline in electroencephalography measurement
Change in Motivation as assessed by Intrinsic Motivation Inventory (IMI) | Before Intervention, Immediately after the end of intervention, at the end of the session
  Intrinsic Motivation Inventory, Self administered. Likert scale of 1-7 (1: not at all true - 4: somewhat true - 7: very true)
Change in Cognitive Load as assessed by National Aeronautics and Space Administration (NASA) (Raw) Task Load Index | Immediately after the end of intervention, At the end of the session
  Self-reported cognitive load during a task, Self-administered National Aeronautics and Space Administration (Raw) Task Load Index (TLX), analog scale mapped from 0 to 100 (Endpoints: Low/High, Good/Poor)
System Usability as assessed by System Usability Scale (SUS) | Immediately after the end of intervention, At the end of the session
  Self reported system usability assessed by System Usability Scale (SUS) Likert scale of 1-5 (Strongly agree to Strongly disagree)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Marchal-Crespo, Prof. Dr., Principal Investigator — University of Bern, ARTORG Center for Biomedical Engineering Research
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be available after publications and it will stay accessible as long as the journal regulation permits.
Access Criteria: Being able to access the journal paper

REFERENCES:
- [Derived] Ozen O, Buetler KA, Marchal-Crespo L. Towards functional robotic training: motor learning of dynamic tasks is enhanced by haptic rendering but hampered by arm weight support. J Neuroeng Rehabil. 2022 Feb 13;19(1):19. doi: 10.1186/s12984-022-00993-w. PMID 35152897